CLINICAL TRIAL: NCT01242943
Title: A PHASE I/II DOSE FINDING AND EFFICACY STUDY OF THE TUMOUR TARGETING HUMAN 131I-L19SIP MONOCLONAL ANTIBODY IN PATIENTS WITH CANCER
Brief Title: Radioimmunotherapy With 131I-L19SIP in Patients With Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: With the determination of the RD and a well established understanding of the safety and tolerability profile, the main endpoints of the study have been met.
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19SIPI131-07/07
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Patients With Cancer
Keywords: I131; L19; antibody; monoclonal; tumour targeting; radioimmunotherapy; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- L19SIP I131 (Experimental): Phase I: Multicentre, open-label, two-step single-arm dose escalation study in sequential cohorts of patients with cancer.
  Phase II: Prospective, open-label, single-arm, multicentre study of 131I-L19SIP, given at the RD as determined in phase I.
  Interventions: Drug: 131I-L19SIP Radioimmunotherapy (RIT)

INTERVENTIONS:
Drug: 131I-L19SIP Radioimmunotherapy (RIT) — Dosimetric evaluation with 131I-L19SIP will be performed to assess eligibility for Radioimmunotherapy.
  Phase I: Patients eligible for Radioimmunotherapy will receive escalating doses of therapeutic 131I-L19SIP administration (intravenously) at the following dosages (expressed in mCi/m2): 111, 139 and 167.

SUMMARY:
The aim of this Study Protocol is to provide a basis for the clinical development of 131I-L19SIP as an anti-cancer therapeutic agent, following the promising results of a Phase I study.

DETAILED DESCRIPTION:
The L19SIP antibody is a fully human antibody, capable of preferential localization around tumor blood vessels while sparing normal tissues. The formation of new blood vessels is a rare event in the adult (exception made for the female reproductive cycle), but is a pathological feature of most aggressive types of cancer. The study aims at determining the therapeutic potential of the L19SIP antibody in SIP format, labelled with the radionuclide 131I, for the treatment of patients with different cancer types. The study follows a Phase I study performed with 131I-L19SIP in over 30 patients with cancer, which has shown an excellent tolerability at radioactive doses as high as 150 mCi and therapeutic benefit for some patients enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cancer, with progressive disease in pre-study period, refractory to conventional standard treatments.
2. Histologically/cytologically confirmed diagnosis of cancer, preferably lung cancer, prostate cancer and colorectal cancer (CRC). At least one measurable (minimum 2.0 cm), non irradiated lesion defined according to modified RECIST criteria, i.e. whenever the measurable disease is restricted to a solitary lesion, its neoplastic nature need not to be confirmed by cytology/histology.
3. ECOG performance status grade 0 or 1.
4. Age ≥18 and ≤ 75 years.
5. Adequate haematological, liver and renal function (haemoglobin ≥ 9 g/dL, absolute neutrophil count (ANC) ≥ 1.50 x 10^9/L; platelets ≥ 100 x 10^9/L, bilirubin within UNL; alkaline phosphatase≤ 2.5 x UNL; ALT, AST ≤ UNL or ≤ 2.5 x UNL in case of liver metastases; albumin ≥ 2.5 g/dL; creatinine ≤ UNL.
6. All acute toxic effects (excluding alopecia) of any prior therapy (including surgery radiation therapy, chemotherapy) must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v.3.0) Grade ≤ 1.
7. Negative serum pregnancy test for females of childbearing potential within 14 days of starting treatment.
8. If of childbearing potential, agreement to use adequate contraceptive methods (e.g. oral contraceptives, condoms, or other adequate barrier controls, intrauterine contraceptive devices, or sterilization) beginning at the screening visit and continuing until 3 months following last treatment with study drug.
9. Evidence of a personally signed and dated IEC-approved Informed Consent indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the study.
10. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.
11. Life expectancy of at least 3 months.
12. Signed and dated informed consent.

Exclusion Criteria:

1. Chemotherapy, radiation, hormonotherapy (with the exception of a gradual titration of LHRH agonists) or immunotherapy or participation in any investigational drug study within 4 weeks of study entry (6 weeks in case of prior nitroureas chemotherapy).
2. Prior radiation dose > 30% of bone marrow volume.
3. Presence of cirrhosis or active hepatitis.
4. Presence of serious cardiac (congestive heart failure, heart insufficiency > grade II NYHA, angina pectoris, myocardial infarction within one year prior to study entry, uncontrolled hypertension or arrhythmia), neurological or psychiatric disorders.
5. Presence of uncontrolled intercurrent illness or any condition which in the judgement of the investigator would place the subject at undue risk or interfere with the results of the study.
6. Recovery from major trauma including surgery within 4 weeks of administration of study treatment.
7. Pregnancy or lactation or unwillingness to use adequate method of birth control.
8. Active infection or incomplete wound healing.
9. Known history of allergy to intravenously administered proteins / peptides / antibodies.
10. Any conditions that in the opinion of the investigator could hamper compliance with the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-11; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Phase I: Maximum tolerated dose (MTD) | 4 weeks
  Establishment of the maximum tolerated dose (MTD) and the recommended dose (RD) for the radiolabelled L19SIP monoclonal antibody.
Phase II: Antitumour activity | 1- 14 months
  Investigation of the antitumour activity of 131I-L19SIP at the RD, in patients with advanced cancer.

SECONDARY OUTCOMES:
Phase I: Study of the variation of radioactivity of 131I in whole blood, at several time intervals (Pharmacokinetics) | 2 days
  Evaluation of the pharmacokinetics of 131IL19SIP.
Phase II: Safety profile | 30 days/ administration
  Determination of the overall safety profile of the iodinated antibody characterized by type, frequency, severity, timing and relationship to study therapy of adverse events and laboratory abnormalities in the first and following cycles in all patients receiving a therapeutic dose.
Phase II: Overall Response Rate (ORR) | 6 and 12 months
  Evaluation of the overall Response Rate (ORR) for all patients having received a therapeutic dose.
Phase II: Progression free survival (PFS) | 6 and 12 months
  Evaluation of the progression free survival (PFS) for all patients having received a therapeutic dose.
Phase II: Survival rate | 6 and 12 months
  Evaluation of the survival rate at 6 and 12 months and overall survival time for all patients having received a therapeutic dose.

CONTACTS AND LOCATIONS:
Overall Officials: Giuliano Mariani, Prof, Principal Investigator — University Hospital Pisa, Italy; Tim Meyer, Dr, Principal Investigator — University College London (UCL) Cancer Institute
Locations (4):
- Italy (3):
  - University Hospital Pisa, Pisa, Tuscany
  - Irst - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori - Meldola (Fc), Meldola
  - Irccs Ospedale Casa Sollievo Della Sofferenza - San Giovanni Rotondo, San Giovanni Rotondo (FG)
- University College London, UCL Cancer Institute, London, United Kingdom